CLINICAL TRIAL: NCT05554510
Title: Prospective Clinical Study of Pulse Oximeter Errors in Hospitalized Patients With Varying Skin Pigmentation
Brief Title: Pulse Oximetry Errors in Hospitalized Patients Across Varying Skin Pigmentation
Acronym: EquiOx
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 22-36553
Record Dates: First submitted 2022-09-09; First posted 2022-09-26 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Hypoxemia; Pulse Oximetry; Skin Pigment
Keywords: Hospitalized Patients
MeSH Terms: conditions — Hypoxia; Pigmentation Disorders | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hospitalized Patients with Arterial Catheters
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — No interventions planned. Observational data collection only.

SUMMARY:
This is a prospective observational study designed to quantify and understand errors in pulse oximetry in hospitalized patients in relation to their skin pigmentation. It is driven by three recent retrospective studies showing missed diagnosis of hypoxemia in patients across a spectrum of skin pigmentation, defined as blood SaO2 <90% when their pulse oximeter reads 92% or greater.

DETAILED DESCRIPTION:
This prospective study will overcome the limitations of earlier retrospective studies using three important study protocols:

1. precise time-matching paired blood gas samples to stable periods of pulse oximeter readings
2. objective quantification of skin pigmentation rather than using documented or self-reported race
3. collection of high quality pulse oximeter tracing data, and identifying potential mediators of discordance of noninvasive and invasive measurements such as low perfusion states.

The primary aim is to quantify the bias in SpO2 measurements across skin pigmentation groups in a real-world setting against the gold standard of invasive measurements of arterial blood oxygen saturation measurements across categories of skin pigmentation. These data are essential to addressing health equity and patient safety for people of all skin pigmentations.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* hospitalized and at high risk of hypoxemia, defined as saturations < 90%,
* patients with arterial line in place for clinical purposes

Exclusion Criteria:

* Profound anemia, defined as hemoglobin < 8 g/dl will preclude blood draws for research purposes
* Known pregnancy
* In custody of law enforcement officials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients at risk for hypoxemia with arterial lines placed for clinical purposes.
Sampling Method: Non-Probability Sample
Enrollment: 757 (Actual)
Dates: Start 2022-08-14 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Pulse Oximetry Errors | Up to 10 simultaneous, paired arterial blood samples and noninvasive pulse oximeter readings obtained during unpredictable qualifying episodes of low oxygen saturation identified by clinically indicated monitoring over a 14-day study period
  Pulse oximeter bias (difference between SpO2 and SaO2)

SECONDARY OUTCOMES:
Occult Hypoxemia Rates | Up to 10 simultaneous, paired arterial blood samples and noninvasive pulse oximeter readings obtained during unpredictable qualifying episodes of low oxygen saturation identified by clinically indicated monitoring over a 14-day study period
  Episodes of arterial blood gas functional saturation <90% with simultaneous pulse oximeter reading >/=92%

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bickler, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General and UCSF Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data without private health information or individual identifiers will be made available via the Open Oximetry Project. De-identified data without sensitive information or identifiers will be shared as outlined in the IRB protocol with the study sponsor, the Unites States Food and Drug Administration.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon study completion, approximately October 2023 and in accordance with any peer-reviewed journal requirements.
Access Criteria: Qualified researchers with appropriate training in Human Subjects Research protocols and without conflicts of interest in data analysis or publication.
URL: https://openoximetry.org/